CLINICAL TRIAL: NCT04824534
Title: Motion Analysis Before and After Surgical Sacroiliac Joint Fusion in Patients With Sacroiliac Joint Dysfunction
Brief Title: Motion Analysis in Sacroiliac Joint Dysfunction
Acronym: MASSIF
Status: Completed | Type: Observational
Sponsor: Zuyderland Medisch Centrum (Other)
Collaborators: Zuyd University of Applied Sciences (Other)
Responsible Party: Principal Investigator, Sem Hermans, Researcher Orthopedic surgery, Zuyderland Medisch Centrum
Other Study IDs: Z2020223
Record Dates: First submitted 2021-03-13; First posted 2021-04-01 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Sacroiliac Joint Dysfunction
Keywords: Movement analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy subjects
  Interventions: Other: Motion analysis
- Healthy subjects matching baseline characteristics with patients
  Interventions: Other: Motion analysis
- Patients with sarociliac joint dysfunction
  Interventions: Other: Motion analysis

INTERVENTIONS:
Other: Motion analysis — Motion analysis is performed in the Motionlab using Vicon systems. Surgery (in case of SI patients) is performed with iFuse implant system for sacroiliac joint fusion

SUMMARY:
Rationale: The sacroiliac joint (SIJ) is increasingly being recognized as a potential cause of chronic low back and buttock pain. The SIJ is affected in 14-22% in patients presenting with this pain. Conservative treatment options include oral analgesic use, physical therapy, radiofrequency denervation and intraarticular steroid injections. When non-surgical treatment remains ineffective, surgical intervention is a reasonable option in the form of minimally invasive sacroiliac joint fusion (MISJF). Recent literature suggests that imbalance and sagittal sacropelvic morphology can occur in patients with SIJ dysfunction.

Using motion analyses, the investigators want to evaluate full movement patterns in SIJ patients. Potentially, changes in these parameters can be observed before and after MISJF surgery.

Objective: To determine spatiotemporal parameters, pelvic obliquity, center of gravity and load capacity in patients suffering from SIJ dysfunction before and after MISJF surgery. Movement parameters will also be determined in healthy individuals to compare with patients suffering from SIJ dysfunction.

Methods: This prospective cohort study will include patients enlisted for MISJF surgery because of SIJ dysfunction. Spatiotemporal parameters, pelvic obliquity, center of gravity and load capacity will be examined before and 3 months after surgery in a professional Motion Lab. Movement parameter of healthy individuals will also be evaluated at the Motion Lab. All data will be analyzed using MATLAB software.

DETAILED DESCRIPTION:
1.2 RATIONALE The sacroiliac joint (SIJ) is an anatomic structure that is increasingly being recognized as a potential cause of chronic low back and buttock pain. The SIJ is affected in 14-22% in patients presenting with this pain.1,2 A wide variability exists in the clinical presentation of SIJ dysfunction, from localized pain around the SIJ to radiating pain into the groin or even the entire lower extremity.3 This sometimes makes it challenging to accurately diagnose SIJ dysfunction during physical examination. Most surgeons palpate the SIJ to determine the level and area of tenderness. There are also several provocative tests, but their reliability is limited.4,5 Currently, diagnostic SIJ intraarticular injection is the benchmark for diagnosing SIJ dysfunction.6 Conservative treatment options include oral analgesic use, physical therapy, radiofrequency denervation and intraarticular steroid injections. 7-11 When non-surgical treatment remains ineffective, minimally invasive sacroiliac joint fusion (MISJF) is a reasonable option.12 Current literature suggests that imbalance and sagittal sacropelvic morphology can occur in patients with SIJ dysfunction.13 Sagittal imbalance and sagittal sacropelvic morphology can in turn lead to compensatory motion in the SIJ, leading to more dysfunction and pain.14 The investigators wonder if changes in spatiotemporal parameters, pelvic obliquity, center of gravity and load capacity can be observed in patients suffering from SIJ dysfunction before and after MISJF surgery with the help of motion analysis. Expectedly, these changes correlate to the clinical condition patients are in

1.3 OBJECTIVES.

This study consists of two different parts, each with different objectives:

1. Process evaluation on measuring movement patterns in the motion lab:

   a. What differences can be detected in spatiotemporal parameters, pelvic obliquity, center of gravity and load capacity between healthy individuals and patients suffering from SI dysfunction?
2. Clinical evaluation of MISJF surgery in patients with SI dysfunction:

   1. What differences can be detected in spatiotemporal parameters, pelvic obliquity, center of gravity and load capacity in patients suffering from SI dysfunction before and after MISJF surgery?
   2. What changes occur in patients suffering from SI dysfunction after MISJF surgery?

2. STUDY DESIGN 2.1 STUDY POPULATION In total 10 patients suffering from SIJ dysfunction with an indication for MISJF, 10 healthy individuals under the age of 25 and 10 healthy individuals matching the demographic characteristics of patients suffering from SI dysfunction will be included. This is a total of 30 individuals.

2.2 INCLUSION CRITERIA

Inclusion criteria for participating clients in the healthy study group:

- Healthy individuals under the age of 25, with no history of SI dysfunction or lower back related illnesses

Inclusion criteria for participating clients in the healthy study group with the same demographic characteristics as the SI dysfunction patients:

- Healthy individuals between the age of 25 and 45, female sex and postpartum with no history of SI dysfunction or lower back related illnesses

Inclusion criteria for the MISJF group:

* The patient is suffering from SIJ dysfunction (uni- or bilateral) because of postpartum pelvic instability or because of Ehlers Danlos syndrome and is enlisted for primary MISJF surgery.
* The patient is mobile enough to perform several tests at the motion lab, needed to obtain spatiotemporal parameters, pelvic obliquity, center of gravity and load capacity.

2.3 EXCLUSION CRITERIA

Exclusion criteria for all participating clients are:

* The individual is not mobile and/or unable to perform tests at the motion lab, needed to obtain spatiotemporal parameters, pelvic obliquity, center of gravity and load capacity.
* Inadequate command of the Dutch language.
* Age under 18 years.

  3. METHODS This prospective study will examine spatiotemporal parameters, pelvic obliquity, center of gravity and load capacity in healthy individuals and patients suffering from SI dysfunction before and after MISJF surgery.

3.1 STUDY PARAMETERS Spatiotemporal parameters, pelvic obliquity, center of gravity and load capacity are the main study parameters and will be determined in the motion lab when walking (gait analysis) and during single leg stance (both sides). Further tests may include straight leg raise while seated and step-ups (both sides).

3.2 STUDY PROCEDURE First, spatiotemporal parameters, pelvic obliquity, center of gravity and load capacity will be determined in 10 healthy individuals under the age of 25. The same parameters will be determined in 10 healthy individuals matching the demographic characteristics of patients suffering from SI dysfunction (female, aged 25 to 45 years and postpartum). Between these two groups potential differences will be evaluated.

In the second part of the study spatiotemporal parameters, pelvic obliquity, center of gravity and load capacity will be determined in patients suffering from SI dysfunction before MISJF surgery. These patients are elected for primary MISJF surgery for SI dysfunction (uni- or bilateral) because of postpartum pelvic instability or because of Ehlers Danlos syndrome. These data will be compared to that of the healthy study group. Spatiotemporal parameters, pelvic obliquity, center of gravity and load capacity will again be measured in the same patients around 3 months after surgery. The pre- and postoperative outcomes will be analyzed and compared. The data from the healthy individuals will be used as reference data in these analyses.

To limit potential biases, the investigators gather extra information from all subjects of the study. Demographic characteristics will be collected, and questionnaires will be conducted on clinical outcomes using visual analog scale (VAS) for pain, Oswestry Disability Index (ODI) for back function and EQ-5D-3L for health-related quality of life.

With regard to the patients suffering from SI dysfunction some additional data on daily activity will be collected. All these patients will carry an activity monitor/accelerometer for the duration of 1 week before and after surgery to determine activity in these patients. Differences before and after surgery will be analyzed in accordance with the spatiotemporal parameters. Finally, the subjects will be asked to give information about the rehabilitation process and physiotherapy (which program, duration, frequency etc.).

4. SAFETY REPORTING During motion analyses all subjects are "visitors" at the motion lab, a liability insurance is in effect during tests. Instructors/researchers are also covered by this insurance. There is no need for additional insurance.

5. STATISTICAL ANALYSIS Demographic baseline characteristics (e.g. age, ASA classification, gender, affected side) of the study participants will be described as descriptives.

5.1 STUDY PARAMETERS The main study parameters are spatiotemporal parameters, pelvic obliquity, center of gravity and load capacity during motion analysis before and after MISJF surgery for the patients suffering from SI dysfunction. These measurements will be collected at the motion lab and analyzed into data to compare different parameters between group differences (healthy versus SI dysfunction e.g.).

Other outcome parameters are change in questionnaires outcome in pain measured in Visual Analogue Scale (VAS) pain score, disability measured using the Oswestry Disability Index (ODI) and change in quality-adjusted life years (QALY) measured with EQ-5D-3L. Analysis of these PROMs will be achieved by linear mixed models to determine the overall effect over time and difference in change of scores at fixed time points and difference in change from baseline/preoperative. Between group differences of baseline scores will also be determined, including data on the rehabilitation process and physiotherapy.

Activity measured by the activity monitors/accelerometers will be a different outcome parameter. Analysis of the activity data will be achieved to determine overall difference in change of scores 3 months after MISJF surgery from baseline/preoperative.

6. ADMINISTRATIVE ASPECTS Demographic baseline characteristics data collection will be carried out using study management software. To protect the privacy of all participants, all collected data will be encoded. The codes that are related to each individual patient are saved in an excel file, which is locked with a password. Only the principal investigator of the specific site will have access to the encoding keys. The outcome parameters from the motion lab will be saved on the software used at HSZ. Data will be exchanged between HSZ and Zuyderland Medical Center using secured emails.

ELIGIBILITY:
Inclusion criteria for participating clients in the healthy study group:

- Healthy individuals under the age of 25, with no history of SI dysfunction or lower back related illnesses

Inclusion criteria for participating clients in the healthy study group with the same demographic characteristics as the SI dysfunction patients:

- Healthy individuals between the age of 25 and 45, female sex and postpartum with no history of SI dysfunction or lower back related illnesses

Inclusion criteria for the MISJF group:

* The patient is suffering from SIJ dysfunction (uni- or bilateral) because of postpartum pelvic instability or because of Ehlers Danlos syndrome and is enlisted for primary MISJF surgery.
* The patient is mobile enough to perform several tests at the motion lab, needed to obtain spatiotemporal parameters, pelvic obliquity, center of gravity and load capacity.

Exclusion criteria for all participating clients are:

* The individual is not mobile and/or unable to perform tests at the motion lab, needed to obtain spatiotemporal parameters, pelvic obliquity, center of gravity and load capacity.
* Inadequate command of the Dutch language.
* Age under 18 years.

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Sacroiliac joint dysfunction mostly effects women.
Study Population: In total 10 patients suffering from SIJ dysfunction with an indication for MISJF, 10 healthy individuals under the age of 25 and 10 healthy individuals matching the demographic characteristics of patients suffering from SI dysfunction will be included. This is a total of 30 individuals.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Change in pelvic obliquity during one leg stance will be collected using VICON Nexus systems. | Before and 3 months after surgery
  measured in mm in 3 different axis
Change in pelvic tilt during one leg stance will be collected using VICON Nexus systems. | Before and 3 months after surgery
  measured in mm in 3 different axis
Change in pelvic obliquity during sit-to-stand task will be collected using VICON Nexus systems. | Before and 3 months after surgery
  measured in mm in 3 different axis
Change in pelvic tilt during sit-to-stand task will be collected using VICON Nexus systems. | Before and 3 months after surgery
  measured in mm in 3 different axis
Change in cadence during gait will be collected using VICON Nexus systems. | Before and 3 months after surgery
  measured in mm in 3 different axis
Change in stride length during gait will be collected using VICON Nexus systems. | Before and 3 months after surgery
  measured in mm in 3 different axis
Change in step width during gait will be collected using VICON Nexus systems. | Before and 3 months after surgery
  measured in mm in 3 different axis
Change in percentage of swing phase during gait will be collected using VICON Nexus systems. | Before and 3 months after surgery
  percentage of total gait
Change in percentage of single support phase during gait will be collected using VICON Nexus systems. | Before and 3 months after surgery
  percentage of total gait
Change in percentage of double support phase during gait will be collected using VICON Nexus systems. | Before and 3 months after surgery
  percentage of total gait
Change in center of gravity during gait will be collected using VICON Nexus systems. | Before and 3 months after surgery
  measured in mm in 3 different axis
Change in center of gravity during one leg stance will be collected using VICON Nexus systems. | Before and 3 months after surgery
  measured in mm in 3 different axis
Change in center of gravity during sit-to-stand tasks will be collected using VICON Nexus systems. | Before and 3 months after surgery
  measured in mm in 3 different axis

SECONDARY OUTCOMES:
Change in Visual Analgogue Scale pain score (0 to 10) | before and 3 months after surgery
Change in disability measured using the Oswestry Disability Index (ODI) | before and 3 months after surgery
Change in quality-adjusted life years (QALY) measured with EQ-5D-5L | before and 3 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Inez Curfs, MD, PhD, Principal Investigator — Zuyderland MC
Locations (1):
- Zuyderland MC, Heerlen, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided